CLINICAL TRIAL: NCT05820126
Title: Cold Versus Room Temperature Storage of Platelets for Bleeding in Hematologic Malignancy - a Pilot Trial
Acronym: CoVeRTS-HM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CoVeRTS-HM
Record Dates: First submitted 2023-04-14; First posted 2023-04-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancy
Keywords: Hematologic malignancies, bleeding, cold-stored platelets
MeSH Terms: conditions — Hematologic Neoplasms; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Single center, Blinded, Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator and participant will both be blinded to the study treatment (whether they receive cold stored vs. room temperature stored platelets). The clinical staff who will administer the platelets and complete the bleeding assessment tool will not be informed of the group assignment. The outcome assessors/adjudication committee will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold-stored platelet concentrate (Experimental): Cold-stored, pathogen-reduced platelet transfusion
  Interventions: Biological: Cold-stored platelet concentrate
- Room temperature-stored platelet concentrate (Other): Room temperature-stored, pathogen reduced platelet transfusion
  Interventions: Biological: Cold-stored platelet concentrate

INTERVENTIONS:
Biological: Cold-stored platelet concentrate — Patients will be transfused a unit of pooled, pathogen reduced platelets that have been stored for >24 hours at 1-6˚C

SUMMARY:
This is a pilot trial to discover the feasibility of recruiting 50 pts over the course of 12 months. The trial is testing the efficacy of using cold-stored vs. room temperature stored (current standard of care) platelets to treat bleeding in persons with hematological disorders and thrombocytopenia.

DETAILED DESCRIPTION:
Patients with hematologic malignancies or marrow aplasia are at increased risk of bleeding. While prophylactic platelet transfusions reduce the risk of bleeding compared with no prophylaxis, a significant risk of bleeding remains, with 43-54% of patients with a hematologic malignancy or marrow aplasia receiving chemotherapy, immunotherapy, or hematopoietic stem cell transplant (HSCT) experiencing WHO grade 2 or higher bleeding [Stanworth et al. NEJM 2013; Gernsheimer et al, Blood 2020]. Improved efficacy of therapeutic platelet transfusions would benefit this patient population. In vitro data suggests that cold-stored platelets have greater hemostatic responsiveness than those stored at room temperature.

This study will evaluate the feasibility of a randomized clinical trial comparing cold- and room temperature storage in patients admitted to hospital with a hematologic malignancy or marrow aplasia. Results will inform estimates of transfusion requirements and changes in bleeding severity for power calculations, inform management of a cold-stored platelet inventory, and will provide data on the use of cold-stored platelets in the Canadian health-care setting.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18) admitted to Malignant Hematology ward with hematologic malignancy or marrow aplasia, this may include patients undergoing chemotherapy, immunotherapy, or hematopoietic stem cell transplant or patients admitted for symptom management.
2. Moderate thrombocytopenia, platelet concentration 10-100 x109/L
3. Platelet transfusion ordered to treat bleeding

Exclusion Criteria:

1. Severe thrombocytopenia (platelet concentration <10 x 109/L)
2. Known platelet refractoriness requiring HLA or HPA selected platelet concentrates
3. International normalized ratio (INR) >2.0
4. Activated partial thromboplastin time (aPTT) >40 seconds
5. Therapeutic anticoagulation (unfractionated heparin, low molecular weight heparin, warfarin, direct oral anticoagulant)
6. Known congenital bleeding disorder
7. History of unprovoked venous thromboembolic disease
8. Transfusion of platelet concentrate for >grade 2 bleeding in preceding 24 hours
9. Order for multiple platelet transfusion at once
10. Refusal of blood transfusion
11. Prior participation in CoVeRTS-HM trial
12. Participation in other clinical trials with interventions that may affect CoVeRTS-HM treatment or outcome
13. Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average Enrollment | 12 months
  1. The primary feasibility outcome is the average number of patients recruited per month.
Enrollment Achieved | 12 months
  50 participants enrolled

SECONDARY OUTCOMES:
Eligible patients consented | 12 months
  Proportion of eligible patients who provide consent
Non-participation | 12 months
  Reasons for non-participation in eligible patients
Protocol Adherance | 12 months
  3. Proportion of patients who complete study procedures and proportion of patients who adhere to the protocol (such as appropriate platelet transfusion, bleeding severity assessment prior to transfusion and at 1-hour, 4 to 6 hours and 18-24 hours after transfusion, platelet count monitoring according to the protocol)
Withdrawal/ Loss to follow up | 12 months
  Rates of withdrawal and loss to follow-up
Expired Cold-platelets | 12 months
  Number of cold-stored platelet concentrates that out-date prior to transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan MAck, MD, Study Chair — McGill University; Alan Tinmouth, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No